CLINICAL TRIAL: NCT00956228
Title: Phase I/II Study of Radioimmunoguided Intensity Modulated Radiotherapy (IMRT) for Prostate Cancer
Brief Title: Study of Radioimmunoguided Intensity Modulated Radiotherapy (IMRT) for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 390-02
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radioimmunoguided IMRT (Experimental): All patients recieved Intensity Modulated Radiotherapy to the prostate with 75.6 Gy in 42 fractions. Additionally, they recieve a concurrent boost to the region of the prostate which enhanced on the prostascint scan to 82 Gy.
  Interventions: Radiation: radioimmuniguided intenstiy modulated radiotherapy

INTERVENTIONS:
Radiation: radioimmuniguided intenstiy modulated radiotherapy — All patients recieved 75.6 Gy in 42 fractions to the prostate and the region of the prostate which enhanced on prostascint scan was simaltaneously boosted to a total dose of 82 Gy

SUMMARY:
The current study involves a novel and aggressive therapeutic approach for patients' prostate cancer. In addition, the investigators propose to administer hormonal therapy to patients with an especially high risk: those with initial Gleason scores of > 6, PSA > 10 ng/ml, T3/T4 primary tumors, and those found to be node positive (N+). The use of hormonal therapy in these specific settings correlates with our current standard of care. IMRT is better able to spare and protect normal tissues from receiving radiation than 3-D conformal RT. The radiotherapy would be followed by continued hormonal therapy for a total of 6 months in those who have one of the following Gleason 7 and PSA 10-20 and as per the previous version of this trial, 1 year similar to that delivered by the EORTC for higher risk patients, (those with initial Gleason scores of > 8, PSA > 20 ng/ml, or T3/T4 tumors). Those found to be N(+) would have the hormonal therapy continued indefinitely or until disease progression occurred in a manner analogous to the Messing et. al. series in prostatectomy patients. The goals are to develop and administer a program of treatment that includes the most recent developments in imaging, integrating data from both the CT scan and the ProstaScint scan to optimize prostate cancer RT. The CT scan will be used for staging and to determine the exact location of the entire prostate which will receive a reasonable dose of RT. The ProstaScint will be used to assess the spread of disease to lymph nodes as well as to determine the exact location of the tumor within the prostate gland. This region will then be boosted to a tumorcidal dose. The investigators then plan to monitor the toxicity and outcome of this treatment. The investigators expect that this program of radioimmunoguided IMRT will likely result in similar or less toxicity and increased cure rates when compared to conventional radiotherapy and standard IMRT programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven prostate cancer
* No evidence of distant metastases (M0) on physical examination, bone scan
* ECOG PS 0,1,2
* Adequate organ function as evidenced by:

  * Hemoglobin > 10.0 gm/dl
  * White blood count > 3000/mcL
  * Platelet count > 90,000/mcL
  * AST < 2x normal
* Age > 18 years
* Patients can not be allergic to Leuprolide or Goserelin if the pretreatment PSA > 20, Gleason Score > 8, T3/4, or N1 disease
* Written informed consent
* We anticipate enrolling at least 50 patients per year, which would bring accrual to projected total of 100 patients in 2 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be assessment of toxicity as well as efficacy as determined by survival rates, freedom from biochemical relapse rates, local control rates, distant failure rates.
The main endpoint of the toxicity component is evaluating how many patients develop grade 3 or greater toxicity.
It is expected between 0 and 9% of patients will have grade 3 or 4 toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States